CLINICAL TRIAL: NCT03612947
Title: Effect of Magnesium Sulfate When Added to TAP Block With Bupivacaine in Patients Undergoing Laparoscopic Cholecystectomy.
Brief Title: TAP Block in Laparoscopic Cholecystectomy.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Seham Mohamed Moeen Ibrahim, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 52018
Record Dates: First submitted 2018-07-19; First posted 2018-08-02 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine +magnesium sulphate (Active Comparator): Ultrasound guided subcostal TAP block will performed on both sides using 20 ml volume (0.25 bupivacaine) plus 150 mg of MgSo4.
  Interventions: Drug: Bupivacaine +magnesium sulphate
- Bupivacaine only (Placebo Comparator): Ultrasound guided subcostal TAP block will performed on both sides using 20 ml volume (0.25 bupivacaine).
  Interventions: Drug: Bupivacaine only

INTERVENTIONS:
Drug: Bupivacaine +magnesium sulphate — Ultrasound guided subcostal TAP block will performed on both sides using 20 ml volume (0.25 bupivacaine) plus 150 mg of MgSo4
  Arms: Bupivacaine +magnesium sulphate
Drug: Bupivacaine only — Ultrasound guided subcostal TAP block will performed on both sides using 20 ml volume (0.25 bupivacaine).
  Arms: Bupivacaine only

SUMMARY:
Ultrasound-guided transversus abdominis plane block is now widely used in abdominal surgery. Recently, magnesium sulphate is used as adjuvant to local anesthetics.

DETAILED DESCRIPTION:
A significant pain experienced by patients after laparoscopic cholecystectomy surgery is required so as to block nociceptive transmission from both the abdominal wall incision, and visceral sites.

Using of opioids can result in significant adverse effects, thus delaying early mobilization of patients.

Ultrasound-guided transversus abdominis plane (TAP) block has been used as a satisfactory approach that provides postoperative analgesia. TAP block is safe; it diminishes or replaces the use of opioids; and it has a lower incidence of adverse effects.

Bupivacaine is a medication used to decrease feeling in a specific area. It is used by injecting it into the area, around a nerve that supplies the area, or into the spinal canal's epidural space. Bupivacaine is indicated for local infiltration, peripheral nerve block, sympathetic nerve block, and epidural and caudal blocks.

Magnesium is the fourth most plentiful cation in our body. It may be worthwhile to further study the role of supplemental magnesium in providing perioperative analgesia, because this is a relatively harmless molecule, is not expensive and also because the biological basis for its potential antinociceptive effect is promising.

Magnesium sulphate (MgSO4), N-methyl-D-aspartate receptor antagonist has the potential to be an ideal adjuvant in TAP block.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age: 18-65 years old) undergoing laparoscopic cholecystectomy.

Exclusion Criteria:

* Patient refusal
* Patients with a history of cardiac, or respiratory diseases ( >ASA III).
* Patients with allergy to amide local anesthetics or medication included in the study.
* Infection at the needle insertion site.
* Pregnancy
* BMI >35
* Drug abusers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
The postoperative pain | The first 24 hours after surgery
  Visual analogue pain score ranging from 0-10 cm where 0 cm
  = no pain and 10 cm = the worst imaginable pain.

SECONDARY OUTCOMES:
Time to first dose of post-operative analgesia | First occurrence during hospitalization (up to 24 hours postoperatively)
  hours
Postoperative nausea and vomiting | The first 24 hours after surgery
  A three-point rating scale (1: no postoperative nausea and vomiting, 2: nausea without vomiting, 3: nausea with vomiting).
postoperative sedation | The first 24 hours after surgery
  Ramsay sedation score as follows: (1) anxious and irritable or dysphoric or both; (2) co-operational, oriented and quiet; (3) responsive to command; (4) asleep, quickly responsive to light tap or loud auditory stimulus; (5) asleep, slowly responsive to light tap or loud auditory stimulus; and (6) asleep, no response to light tap or loud auditory stimulus.
Patient satisfaction | At 24 hours after surgery
  Patient satisfaction score ranged from 0-100 points; with 0 indicating the worst level of satisfaction and 100 indicating the best level of satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Assuit University, Asyut, Asyut Governorate, Egypt